CLINICAL TRIAL: NCT02885038
Title: Analyse de l'Effet Des caractéristiques de concentrés Plaquettaires Sur le Rendement Transfusionnel Chez Les Patients Ayant Une hémopathie Maligne et bénéficiant de Transfusions Plaquettaires à Titre Prophylactique
Brief Title: Effect of Product Related Factors on Platelet Concentrate Transfusion Response in Patients With Hematologic Malignacies
Acronym: TCP
Status: Completed | Type: Observational
Sponsor: Etablissement Français du Sang (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: CPP14/05; DR-2015-392 (Other: French Data Protection Authority)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2016-09

CONDITIONS: Lymphoma; Multiple Myeloma; Lymphocytic Leukemia; Hodgkin Disease
Keywords: Platelet Transfusion
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Leukemia, Lymphoid; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Platelet concentrate transfusion

SUMMARY:
Platelet concentrates (PCs) characteristics, such as storage duration, ABO compatibility, dose and source, may have an impact on transfusion responses and outcomes. Because of the relative scarcity of PCs the selection of a specific PC for issue to the patient remains a challenging process. Regulatory agencies do not fully address these characteristics in their recommendations for prophylactic transfusions.

The aim of the study was to analyse the effect of product-related factors in a real life setting, in order to determine which ones are the most relevant when selecting PCs for patients in prophylactic conditions. Two different endpoints are studied: the corrected count increment and the platelet transfusion time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in the hematology department between January 2001 and December 2012
* Hematologic malignancy
* At least one platelet transfusion (with platelet count ≤ 25 G/L)
* Age 18 and over at time of first transfusion

Exclusion Criteria:

* More than one hematologic malignancy
* Non-malignant haematological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with hematologic malignancies treated at the university hospital of Besançon who received at least one prophylactic platelet transfusion
Sampling Method: Non-Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Corrected count increment | 24 hours post transfusion
  Platelet increment corrected for platelet dose and body surface area

SECONDARY OUTCOMES:
Transfusion interval | 7 days
  Time interval to following platelet transfusion in days

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BARDIAUX, MD, Principal Investigator — Etablissement Français du Sang

IPD SHARING:
Plan to Share IPD: Undecided